CLINICAL TRIAL: NCT06218979
Title: KF2022#3-tutkimus: Teen Ja Kolajuoman Vaikutus Risperidoni-oraaliliuoksen Imeytymiseen
Brief Title: KF2022#3-trial: Effect of Tea and Cola Beverage on Absorption of Risperidone Oral Solution
Acronym: KF2022#3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Janne Backman, Professor, head physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KF2022#3
Record Dates: First submitted 2023-12-04; First posted 2024-01-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Psychosis; Food-drug Interaction
MeSH Terms: conditions — Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control phase (Placebo Comparator): Study drug dose (1 mg risperidone) and 250 ml of water at 8:00 a.m., and 250 ml of water at 8:30 a.m.
  Interventions: Drug: Risperidone oral solution
- Tea phase (Active Comparator): Study drug dose (1 mg risperidone) and 250 ml of tea at 8:00 a.m., and 250 ml of tea at 8:30 a.m.
  Interventions: Drug: Risperidone oral solution
- Cola beverage phase (Active Comparator): Study drug dose (1 mg risperidone) and 250 ml cola drink at 8:00 a.m., and 250 ml cola beverage at 8:30 a.m.
  Interventions: Drug: Risperidone oral solution

INTERVENTIONS:
Drug: Risperidone oral solution — See arm/group descriptions
  Other Names: Twinings English Breakfast tea; Pepsi Max beverage

SUMMARY:
Risperidone is widely used in the treatment of schizophrenia, bipolar disorder, and aggression associated with moderate or severe Alzheimer's dementia. In vitro studies have shown that constituents of tea and cola beverages can result in insoluble complex formation with risperidone, potentially reducing risperidone oral absorption. The purpose of this study is to investigate the effect of tea and cola beverage on the pharmacokinetics of risperidone oral solution.

In an open three-phase, randomized, crossover study with 12 healthy volunteers, the subjects will receive a 1 mg dose of risperidone oral solution with either water, tea or cola beverage. Blood samples will be collected and risperidone's pharmacokinetics will be monitored up to 48 hours postdose. Primary endpoint is area under the plasma concentration-time curve of risperidone.

Recruitment starting date is December 4, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-45
* Healthy
* Systolic blood pressure ≥110 mmHg
* Heart rate ≥ 50/min
* Normal ECG
* Accepted results from laboratory tests (blood haemoglobin, basic blood count and blood platelets, alanine aminotransferase, alkaline phosphatase, glutamyl transferase, creatinine, plasma potassium and sodium). Negative pregnancy test result (serum human chorionic gonadotropin) for women.

Exclusion Criteria:

* Significant disease
* Mood disorder or suicidality
* Smoking
* Using oral contraception pills or other regular medication
* Pregnancy (current or planned) or nursing
* Participation in any other studies involving investigational or marketed drug products within three months prior to the entry into this study
* Donation of blood within three months prior to the entry into this study
* Significant overweight / small or hard-to-find veins
* BMI < 18.5 kg/m2
* Insufficient Finnish language skills

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve of risperidone | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone

SECONDARY OUTCOMES:
Peak plasma concentration for both risperidone and its metabolites | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone
Half-life for both risperidone and its metabolites | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone
Time to peak plasma concentration for both risperidone and its metabolites | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone
Fractional areas under concentration-time curve (AUC) for both risperidone and its metabolites | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone
Areas under concentration-time curve (AUC) for risperidone metabolites | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone
CYP2D6 activity biomarkers (solanidine and its metabolites) | Prior to and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 11, 24, and 48 hours after administration of risperidone

CONTACTS AND LOCATIONS:
Overall Officials: Janne Backman, MD, PhD, Principal Investigator — Professor, Head physician
Locations (1):
- Department of Clinical Pharmacology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No